CLINICAL TRIAL: NCT00843804
Title: Prospective Surveillance for Nosocomial Infections and Catheter-related Thrombotic Events in Pediatric Patients
Brief Title: Surveillance for Nosocomial Infections in Pediatric Cancer Patients
Acronym: Oncoped2006
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Arne Simon (MD, PhD), Childrens Hospital medical Center, University of Bonn
Other Study IDs: 03/07
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2009-02

CONDITIONS: Nosocomial Infections; Bloodstream Infection; Invasive Aspergillosis
Keywords: nosocomial infection; bloodstream infection; central venous catheter; invasive Aspergillosis; Clostridium difficile associated disease
MeSH Terms: conditions — Cross Infection; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood culture isolates
Oversight: Data Monitoring Committee: No

SUMMARY:
The Oncoped 2006 study implements a multicenter prospective surveillance module for nosocomial infections in pediatric cancer patients.

DETAILED DESCRIPTION:
Type of study:

Prospective multicenter surveillance study referring to file data collected routinely during the management of infectious and thrombotic complications in high risk pediatric cancer patients.

Primary aims of the Oncoped 2006 Study

1. To describe the epidemiology of selected nosocomial infections in pediatric cancer patients as well on the unit level as in a reference database of cumulative data from a prospective multicenter surveillance perspective.
2. To allow the participating institution

   * to compare its own results with other centers and with the reference database (median and 75. percentile).
   * to reduce the incidence density of nosocomial infections and the incidence rate of catheter-associated infections in pediatric cancer patients.
3. To promote patient's safety by means of quality assurance and a reduction of nosocomial infections.
4. To describe objective outcome variables related to the documented NI events (mortality, duration of hospitalization, need for intensive care, need for surgical interventions)
5. To intensify the practical collaboration of the health care team with infection control personnel and infectious disease specialists in this clinical context.
6. To describe the distribution of bacterial pathogens of blood stream infections and to determine the sensitivity (minimal inhibitory concentration) of bacterial pathogens detected in blood cultures to first and second line antimicrobial agents in this high risk population with a standardized method (central reference laboratory).
7. To detect bacterial isolates with emerging types of antimicrobial resistance.
8. To describe the therapeutic use of antibacterial and antifungal agents in pediatric cancer patients related to nosocomial infections.
9. To describe the incidence and incidence density of invasive Aspergillosis in pediatric cancer patients.
10. To describe the clinical impact of common and emerging viral respiratory pathogens (RSV, Influenza, hMPV, hCoV, hBoV) in pediatric cancer patients with nosocomial lower respiratory tract infection (central reference laboratory for emerging viral pathogens).
11. What is the incidence and incidence rate (per 1000 catheter utilization days) of thrombotic events in pediatric cancer patients and in patients with hemophilia, who have a CVAD in use?
12. How many of the children with an event do have congenital risk factors (thrombophilia)?
13. What are the objective outcome parameters in this population considering antithrombotic treatment (at the discretion of the attending physicians)?

ELIGIBILITY:
Inclusion Criteria:

* pediatric cancer patients receiving inpatient treatment with chemotherapy, -
* radiotherapy or stem cell transplantation

Exclusion Criteria:

* no informed consent
* no inpatient treatment

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with cancer during intensive induction / reinduction treatment (including conventional chemotherapy, radiotherapy and stem cell transplantation).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-03; Study Completion 2010-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Arne Simon, MD, Principal Investigator — Children's Hospital Medical Center, University of Bonn, Germany; Roland Ammann, MD, Study Director — Children's Hosptial, Bern, Switzerland; Hans-Jürgen Lawas, MD, Study Chair — Children's Hospital Medical Center, Düsseldorf, Germany
Locations (1):
- Children's Hospital, Pediatric Oncology UNit, Bern, Switzerland

REFERENCES:
- [Background] Simon A, Fleischhack G, Hasan C, Bode U, Engelhart S, Kramer MH. Surveillance for nosocomial and central line-related infections among pediatric hematology-oncology patients. Infect Control Hosp Epidemiol. 2000 Sep;21(9):592-6. doi: 10.1086/501809. PMID 11001263
- [Background] Simon A, Bode U, Fleischhack G, Kramer M. Surveillance of nosocomial infections in pediatric cancer patients. Am J Infect Control. 2005 Dec;33(10):611. doi: 10.1016/j.ajic.2005.09.005. No abstract available. PMID 16330311
- [Background] Simon A, Fleischhack G, Wiszniewsky G, Hasan C, Bode U, Kramer MH. Influence of prolonged use of intravenous administration sets in paediatric cancer patients on CVAD-related bloodstream infection rates and hospital resources. Infection. 2006 Oct;34(5):258-63. doi: 10.1007/s15010-006-5646-y. PMID 17033749
- [Background] Simon A, Groger N, Wilkesmann A, Hasan C, Wiszniewsky G, Engelhart S, Kramer MH, Bode U, Ammann RA, Fleischhack G. Restricted use of glycopeptides in paediatric cancer patients with fever and neutropenia. Int J Antimicrob Agents. 2006 Nov;28(5):417-22. doi: 10.1016/j.ijantimicag.2006.08.007. Epub 2006 Oct 12. PMID 17046210
- [Background] Simon A, Besuden M, Vezmar S, Hasan C, Lampe D, Kreutzberg S, Glasmacher A, Bode U, Fleischhack G. Itraconazole prophylaxis in pediatric cancer patients receiving conventional chemotherapy or autologous stem cell transplants. Support Care Cancer. 2007 Feb;15(2):213-20. doi: 10.1007/s00520-006-0125-7. Epub 2006 Aug 30. PMID 16944217